CLINICAL TRIAL: NCT01128257
Title: Controllability and Real Life Efficacy of Bonviva 3 mg iv Quarterly vs. Oral Alendronate Generics
Brief Title: A Study of Ibandronate [Bonviva/Boniva] and Alendronate in Female Patients With Post-Menopausal Osteoporosis
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML22927
Record Dates: First submitted 2010-05-03; First posted 2010-05-21 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Postmenopausal Osteoporosis
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Alendronate; Ibandronic Acid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- 1
  Interventions: Drug: ibandronate [Bonviva/Boniva]
- 2
  Interventions: Drug: alendronate

INTERVENTIONS:
Drug: alendronate — As prescribed by physician
  Groups: 2
Drug: ibandronate [Bonviva/Boniva] — As prescribed by physician
  Groups: 1

SUMMARY:
This observational study will assess the compliance and persistence of patients, real life efficacy and safety of intravenously quarterly administered 3 mg ibandronate [Bonviva/Boniva] in comparison to oral alendronate generics in female patients with post-menopausal osteoporosis. The anticipated time of assessment is 12 months. The target sample size is 5000-7000 patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 55 years of age
* Postmenopausal osteoporosis
* Patients who are in the opinion of the physician eligible to participate in this study

Exclusion Criteria:

* N/A

Min Age: 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female post-menopausal patients over the age of 55 years
Sampling Method: Probability Sample
Enrollment: 6054 (Actual)
Dates: Start 2010-04; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Assessment of compliance and persistence of Bonviva therapy: Number of prescriptions, number of applied injections, number of taken oral medication, continuation and duration of treatment | 12 months

SECONDARY OUTCOMES:
Pain intensity and reduction in use of analgesics | 12 months
Quality of life and patients satisfaction | 12 months
Degree of patient's mobility | 12 months
Incidence of new osteoporotic fractures | 12 months
Controllability and management of therapy by the physician | 12 months
Patient baseline characteristics | 12 months
User friendliness | 12 months
Safety: AEs and SAEs | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Marburg, Germany